CLINICAL TRIAL: NCT04810936
Title: A Randomized Controlled Trial of an Early Oral Nutritional Supplements Intervention Versus a Conventional Nutritional Intervention in Patients With Locally Advanced Nasopharyngeal Carcinoma Undergoing Concurrent Chemoradiotherapy
Brief Title: Early Nutritional Intervention in NPC Patients Undergoing Concurrent Chemoradiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, YI PAN, Prof., Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GDREC2018296H(R1)
Record Dates: First submitted 2021-03-14; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Malnutrition; Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; malnutrition; Early nutritional intervention; chemoradiotherapy
MeSH Terms: conditions — Malnutrition; Nasopharyngeal Carcinoma | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early ONS intervention group (Experimental): Patients in early ONS intervention group will receive nutritional counseling (follow-up visits once a week during radiotherapy and at the 1st and 3rd months after radiotherapy) and ONS intervention in the beginning of radiotherapy. The ONS is prescribed to increase oral intake of patients and to ensure total energy supply is more than 30 kcal/kg/day and protein intake more than 1.2 g/kg/day.
  Interventions: Dietary Supplement: oral nutritional supplements
- Standard nutrition intervention group (No Intervention): Patients in standard nutrition intervention group will receive nutritional counseling (follow-up visits once a week during radiotherapy and at the 1st and 3rd months after radiotherapy).

INTERVENTIONS:
Dietary Supplement: oral nutritional supplements — Oral nutritional supplements is usually administrated to improve nutritional status in cancer patients.
  Arms: Early ONS intervention group

SUMMARY:
This single center, open-label, randomized controlled clinical trial was designed to investigate whether early nutritional intervention with oral nutrition supplements in patients with nasopharyngeal carcinoma undergoing chemoradiotherapy will improve nutritional status, quality of life and treatment tolerance.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the standard treatment for locally advanced nasopharyngeal carcinoma (NPC). During chemoradiotherapy, malnutrition is present in 44-88% patients which is associated with adverse clinical outcomes. Although patients receive conventional nutritional intervention recommended by The European Society for Clinical Nutrition and Metabolism guidelines, there are still 35% NPC patients suffering from malnutrition during chemoradiotherapy.

Recent studies have shown that early nutritional intervention before radiotherapy reduced the prevalence of malnutrition. However, there are few randomized controlled clinical studies comparing early oral nutritional supplements (ONS) intervention to conventional nutritional intervention in NPC patients undergoing chemoradiotherapy.

This single center, open-label, randomized controlled clinical trial was designed to investigate whether early ONS intervention compared to conventional nutritional intervention improves nutritional status, treatment tolerance and quality of life, and decreases the incidence of grade 3-4 treatment related side-effects in NPC patients undergoing chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed nasopharyngeal carcinoma (NPC).
* The clinical stage of NPC is T1-4 N1-3 M0 (AJCC 7th edition).
* Planned to receive concurrent chemoradiotherapy with intensity-modulated radiation therapy (IMRT).
* Age ≥ 18 years and < 75 years.
* Performance status (PS) score 0-1.
* NRS2002<3 .
* Blood regular test should be satisfied the following conditions: white blood cell count ≥3.5×109/L， Neutrophil count ≥1.5×109/L，platelet count ≥100×109/L，hemoglobin ≥10g/L
* Liver and kidney functions test should be satisfied the following conditions: aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2.5 times the upper limit of normal value, bilirubin < 1.2 times the upper limit of normal value, creatinine < 1.2 times the upper limit of normal value, and alkaline phosphatase < 5 times the upper limit of normal value.
* Could complete required oral nutrition, questionnaire survey and follow-up.
* Signed informed consent voluntarily.

Exclusion Criteria:

* Had a history of head and neck radiotherapy.
* Known allergic reaction to any component of ONS, or severe allergic constitution.
* With any unstable systemic disease (such as uncontrolled infectious diseases, uncontrolled hypertension, uncontrolled metabolic diseases and so on).
* Serious cardiovascular diseases in 6 months (such as Congestive heart failure and myocardial infarction).
* Pregnancy and lactation.
* Other conditions that the investigators consider as inappropriate for enrolling into this study.
* Has a history of malignant tumors in 5 years, except for tumors that have been cured only by surgery and with a disease free survival for five years, cured basal cell carcinoma of skin and cured carcinoma in situ of the cervix.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who lose >5% of initial body weight | 7 weeks
  Assess body weight at the end of radiotherapy (the weight at the end of radiotherapy - the weight at the beginning of radiotherapy) / the weight at the beginning of radiotherapy *100 %.

SECONDARY OUTCOMES:
Weight loss at the last day of radiotherapy | 7 weeks
  The changes of weight at the last day of radiotherapy
Weight loss at the end of 4th week | 11 weeks
  The changes of weight at the end of 4th week
Patient-generated Subjective Global Assessment (PG-SGA) at the end of the 2nd week, 4th week, the last day of radiotherapy and 1 month after radiotherapy | 11 weeks
  PG-SGA at the end of the 2nd week, 4th week, the last day of radiotherapy and 1 month after radiotherapy
Incidence of radiation induced grade 3-4 mucositis (CTCAE 4.03) at the end of 4th week and the last day of radiotherapy | 7 weeks
  Incidence of radiation induced grade 3-4 mucositis at the end of 4th week and the last day of radiotherapy
Incidence of any grade 3-4 side-effect (CTCAE 4.03). | 7 weeks
  Incidence of any grade 3-4 side-effect induced by radiotherapy or chemotherapy during chemoradiotherapy
Incidence of prolonged radiation treatment time caused by side-effects | 7 weeks
  Incidence of prolonged radiation treatment time caused by chemoradiation related side-effects. Prolonged radiation treatment time is defined as the overall treatment time is longer than plan
Days prolonged more than planed treatment time caused by side-effects | 7 weeks
  Days prolonged more than planed treatment time caused by chemoradiation related side-effects
Incidence of unplanned hospitalization in 3 months after radiation | 5 months
  Incidence of unplanned hospitalization in 3 months after radiation. Unplanned hospitalization is defined as hospitalization caused by chemoradiotherapy related side effects
The changes of QOL-C30 at the end of radiation, the 1st and the 3rd month after radiation as compared with the beginning of radiation | 5 months
  The changes of QOL-C30 at the end of radiation, the 1st and the 3rd month after radiation as compared with the beginning of radiation
The treatment time of parenteral nutrition (PN) treatment | 5 months
  PN should be started if enteral nutrition (EN) is anticipated (60% of estimated energy expenditure) for more than 10 days. The treatment time of PN should be recorded
The changes of EORTC Quality of LifeQuestionnaire (QLQ)-H&N35 at the end of radiation, the 1st and the 3rd month after radiation as compared with the beginning of radiation | 5 months
  The changes of EORTC Quality of LifeQuestionnaire (QLQ)-H&N35 at the end of radiation, the 1st and the 3rd month after radiation as compared with the beginning of radiation

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided